# Psychological treatment of hypersexuality: a clinical trial with Acceptance and Commitment Therapy

ID: CIPI/21/003

Document date: 8<sup>th</sup> February 2021

IP: Francisco Montesinos, Ph.D.

Informed consent form

# INFORMED CONSENT FORM TO PARTICIPATE IN THE RESEARCH: "PSYCHOLOGICAL FLEXIBILITY PROGRAM FOR THE IMPROVEMENT OF SEXUAL HEALTH"

We would like to invite you to participate in this research developed by a team of professors from the Department of Psychology of the European University of Madrid. The program is aimed at Spanish-speaking people of legal age who wish to improve the control of their sexual impulses and have a fuller life.

Participate only if you wish to do so. If you choose not to participate, it will not be any inconvenience for you. Before deciding if you want to participate, it is important that you understand why this research is being done and what your participation will entail. Take your time to read the following information and ask us if something is unclear or if you want more information.

#### WHAT DOES IS THIS STUDY ABOUT?

The objective is to evaluate the effectiveness of a psychological flexibility program that aims at helping people who do not feel satisfied with their sexuality and, in particular, who want to improve the control of their sexual impulses.

The results obtained will help us create effective intervention protocols. In addition, participation may be helpful in handling other situations where you may struggle.

#### WHAT WILL I BE ASKED TO DO IF I PARTICIPATE IN THIS STUDY?

- You will have the possibility to participate in a free individual psychological intervention to promote psychological flexibility led by a psychologist/ researcher.
- We will ask you to attend one evaluation session and eight online intervention sessions through Skype or another equivalent platform.
- The sessions will be recorded for future analysis.
- You will have to complete a few questionnaires at three different times: at the beginning
  of your participation, at the end of the program and after three months.

#### WILL MY INFORMATION BE KEPT PRIVATE?

Your answers will be confidential. We will not collect any identifying information. The entire research process will be carried out guaranteeing the anonymity of the participants, and the voluntariness of the participation. The data will be treated in accordance with Royal Decree-Law 5/2018, of July 27, on urgent measures for the adaptation of Spanish Law to European Union regulations on data protection.

The data collected will only be accessible to the study researchers. When the results are reported in congresses or publications, only group summary data will be included, and it will not be possible to identify specific responses.

#### WHO CAN I TALK TO IF I HAVE QUESTIONS ABOUT THIS STUDY?

If you need any further clarification, you can contact the researchers of this study:

- Francisco Montesinos, Department of Psychology of the European University, on phone
   +34912115108 or using the email francisco.montesinos@universidadeuropea.es
- Marta Ortega Otero, using the email marta.ortega@universidadeuropea.es

### WHAT ARE MY RIGHTS AS A RESEARCH STUDY VOLUNTEER?

Your participation is entirely voluntary. There will be no penalty for you if you choose not to participate.

## WHAT DOES IT MEAN THAT I GIVE MY CONSENT?

- That you have understood the information provided in this questionnaire and that you
  are willing to participate in the study.
- That you have had the opportunity to ask questions to the researcher and discuss any concerns.
- That the researcher responded to your questions and concerns appropriately.

#### Declaration of consent

#### I declare:

- 1. That I am of legal age and that I have read and understood all the oral and written information in relation to the participation in the aforementioned project.
- 2. I have had the opportunity to discuss and ask about this information and I have received the appropriate answers from one of the members of the research team in charge of this study.
- 3. I have been assured that the data is confidential.
- 4. I voluntarily consent to participate in this study by attending the training program and completing the questionnaires at different times in time.
- 5. I commit to do my best to complete the treatment and attend the nine sessions (one evaluation and eight intervention), and to notify the therapist at least 24 hours in advance in the event of not being able to attend an appointment.
- 6. I voluntarily give consent and I am aware that I am free to withdraw from the study at any time during the study, for any reason and without having to give any explanation.

| l, | , with ID number |
|---|---|
| and date of birth | I consent to my participation in the study in the term |
| expressed above. | |
| In Madrid, on the of | of 202_ |

Signature